CLINICAL TRIAL: NCT03782831
Title: Transarterial Chemoembolization Plus Programmed Cell Death Protein-1 Antibody Versus Transarterial Chemoembolization Alone for Unresectable Hepatocellular Carcinoma
Brief Title: TACE Plus PD-1 Antibody vs TACE Alone for Unresectable HCC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Sun Yat-sen University (Other)
Collaborators: Kaiping Central Hospital (Other); Guangzhou No.12 People's Hospital (Other Government)
Responsible Party: Principal Investigator, Shi Ming, Proffessor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HCC-S066
Record Dates: First submitted 2018-12-19; First posted 2018-12-20 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2018-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Programmed cell death protein-1 antibody; Transarterial chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — spartalizumab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TACE plus PD-1 antibody (Experimental): Patients received hepatic intra-arterial infusion with lipiodol mixed with chemotherapy drugs (EADM, lobaplatin, and MMC), and embolization with polyvinyl alcohol particles (PVA) on demand. In addition, patients received 3mg/kg PD-1 antibody intravenously every 2 weeks up to documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent.
  Interventions: Procedure: TACE; Drug: PD-1 antibody
- TACE alone (Active Comparator): Patients received hepatic intra-arterial infusion with lipiodol mixed with hemotherapy drugs (EADM, lobaplatin, and MMC), and embolization with polyvinyl alcohol particles (PVA) on demand. In addition, patients received placebos intravenously every 2 weeks
  Interventions: Procedure: TACE; Drug: Placebos

INTERVENTIONS:
Procedure: TACE — Hepatic intra-arterial infusion with lipiodol mixed with chemotherapy drugs (EADM, lobaplatin, and MMC), and embolization with polyvinyl alcohol particles (PVA).
Drug: PD-1 antibody — 3mg/kg intravenously every 2 weeks
  Arms: TACE plus PD-1 antibody
Drug: Placebos — intravenous injection every 2 weeks
  Other Names: normal saline
  Arms: TACE alone

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of transarterial chemoembolization (TACE) combined with programmed cell death protein-1 (PD-1) antibody compared with TACE Alone in patients with unresectable hepatocellular carcinoma (HCC)

DETAILED DESCRIPTION:
Transarterial chemoembolization (TACE) is the first-line treatment for patients with unrestable hepatocellular carcinoma (HCC) at intermediate-stage. Programmed cell death protein-1 (PD-1) antibody is effective and safe for advanced HCC. No study has compared the efficacy and safety of TACE plus PD-1 antibody and TACE alone. Thus, the investigators carried out this prospective randomized control study to find out it.

ELIGIBILITY:
Inclusion Criteria:

* KPS≥70;
* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL), simultaneously staged as BCLC A or BCLC B based on Barcelona Clinic Liver Cancer staging system.
* Patients must have at least one tumor lesion that can be accurately measured;
* Diagnosed as unresectable with consensus by the panel of liver surgery experts;
* Re commanded treated by TACE with consensus by the panel of liver MDT;
* No past history of TACE, chemotherapy or molecule-targeted treatment;
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Meet the following laboratory parameters:(a) Platelet count ≥ 75,000/μL; (b)Hemoglobin ≥ 8.5 g/dL;(c) Total bilirubin ≤ 30mmol/L;(d) Serum albumin

  ≥ 32 g/L;(e) ASL and AST ≤ 6 x upper limit of normal;(f) Serum creatinine

  ≤ 1.5 x upper limit of normal;(g) INR > 2.3 or PT/APTT within normal limits; (h) Absolute neutrophil count (ANC) >1,500/mm3;
* Ability to understand the protocol and to agree to and sign a written informed consent document.

Exclusion Criteria:

* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known of serious heart disease which can nor endure the treatment such as cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Evidence of bleeding diathesis.
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug
* Serious non-healing wound, ulcer, or bone fracture
* Known central nervous system tumors including metastatic brain disease
* Poor compliance that can not comply with the course of treatment and follow up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 12 months
  PFS was defined as the time from the date of randomization to the date of first documentation of disease progression based on modified Response Evaluation Criteria in Solid Tumors (mRECIST), or date of death, whichever occurred first.

SECONDARY OUTCOMES:
Overall Survival (OS) | 12 months
  OS was defined as the duration from the date of randomization until the date of death from any cause. Participants who were lost to follow-up were censored at the last date the participant was known to be alive, and participants who remained alive were censored at the time of data cutoff.
Objective Response Rate (ORR) | 12 months
  ORR was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) based on mRECIST. CR was defined as disappearance of any intratumoral arterial enhancement in all target lesions. PR was defined as at least a 30% decrease in the sum of diameters of viable (enhancement of arterial phase) target lesions taking as reference to the baseline sum of the diameters of target lesions.
Adverse Events | 12 months
  Number of adverse events. Postoperative adverse events were graded based on CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, MD, Principal Investigator — Sun Yat-sen University
Locations (3):
- China (3):
  - Cancer Center Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou Twelfth People's Hospital, Guangzhou, Guangdong
  - Kaiping Central Hospital, Kaiping, Guangdong